CLINICAL TRIAL: NCT03225521
Title: HeartSteps: a Just-in-Time Adaptive Intervention for Increasing Physical Activity Amongst Sedentary Adults.
Brief Title: A Micro-randomized Trial of HeartSteps, an mHealth Intervention for Increasing Physical Activity
Acronym: HS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HUM00103127; 5R01HL125440 (NIH)
Record Dates: First submitted 2017-07-19; First posted 2017-07-21 (Actual); Last update posted 2018-10-25 (Actual); Status verified 2018-10

CONDITIONS: Physical Activity
Keywords: Physical Activity; Mobile Health; Self Monitoring; Wearable Sensors; Tailored Health Communication; Implementation Intentions; Mobile Apps; Anti-Sedentary Behavior; Opportunistic Physical Activity; Health Belief Model
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: Each participant-time point is randomized between intervention or no intervention (delivery of a contextually tailored activity suggestion or no suggestion; planning or no planning)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HeartSteps intervention (Experimental): For activity suggestions, at each available decision time, each participant is randomly assigned to either receive an activity suggestion or not. The randomization probability is 0.6 for receiving a message and 0.4 for not receiving a message.
  For activity planning, at each decision point, the participant is randomized to either receive evening planning or not at that decision time. The randomization probability for receiving planning is 0.5, and 0.5 for not receiving planning.
  Interventions: Behavioral: HeartSteps: A just-in-time adaptive intervention for increasing physical activity amongst sedentary adults.

INTERVENTIONS:
Behavioral: HeartSteps: A just-in-time adaptive intervention for increasing physical activity amongst sedentary adults. — HeartSteps is an Android-based mHealth intervention that contains two main intervention components: contextually-tailored suggestions for activity and planning of the next day's activity. Activity suggestions provide individuals with actionable suggestions for how they can be active in their current context. Delivered suggestions are tailored based on time of day, user's location, day of the week (weekend/weekday), and weather. HeartSteps can deliver a user activity suggestions up to five times a day. Evening planning asks users to create or choose a plan of how they will be active on the following day. Planning can be delivered once a day, in the evening.

SUMMARY:
The aim of this research is to evaluate the efficacy of contextually tailored activity suggestions and activity planning for increasing physical activity among sedentary adults.

DETAILED DESCRIPTION:
Physical activity is a key behavioral strategy for prevention of non-communicable diseases such as diabetes and heart disease. Mobile health (mHealth) interventions have shown promise for supporting physical activity adoption and maintenance in ways that are highly acceptable to users, scalable, and cost-efficient. This study examines two intervention strategies-contextually tailored activity suggestions and daily planning of the activity for the next day-that a mobile health intervention can use to encourage physical activity in sedentary adults.

Study participants use HeartSteps, an mHealth physical intervention developed by the research team, in their daily lives for six weeks. Over the course of the study both of the HeartSteps intervention components-contextually-tailored activity suggestions and activity planning-are micro-randomized for each participant on each of the day of the study, in order the effects on physical activity of each component separately and how those effects change over time.

The primary hypothesis for suggestions is that providing a contextually tailored activity suggestion increases participant step count over the subsequent 30 minutes following message delivery.

The first secondary hypothesis for suggestions is that the proximal effect of the contextually tailored activity suggestions on the subsequent 30-minute step count will decrease with duration in the study.

The primary hypothesis for planning is that receiving evening planning will increase step count on the following day.

The primary analyses will use the methods developed in Boruvka et al. (2017). The primary longitudinal outcome for activity suggestions will be the log of the step count in the 30 minutes subsequent to decision points. The log of the step count in the 30 minutes prior to randomization will be included as a control variable. The primary longitudinal outcome for planning will be the square root of the step count on the day following the randomization of planning treatment.

All missing but "available" minute-by-minute step counts from the wrist band will be imputed as 0. See "Allocation" section for the definition of availability. Sensitivity analyses using step counts from the mobile phone (secondary data source) will be conducted.

ELIGIBILITY:
Inclusion Criteria:

* English speakers,
* between 18 and 60 years of age,
* could walk for exercise without discomfort, and
* either had a full-time daytime job or a regular schedule outside the home (e.g., students)
* have a personal phone running Android 5.0 or higher or willing to use a study-provided phone as their primary phone for the duration of the study.

Exclusion Criteria:

* Need medical supervision to exercise
* Currently using an activity tracker (e.g., FitBit)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2015-07-18 (Actual); Primary Completion 2016-02-01 (Actual); Study Completion 2016-02-01 (Actual)

PRIMARY OUTCOMES:
30 minute step count | 30 minutes
  30-minute window after each available decision point
Daily step count | 24 hour day
  Daily step count on the day following treatment

SECONDARY OUTCOMES:
Thumbs up/down | 30-minute window while message is available
  User ratings of message usefulness (thumbs up/thumbs down rating)

IPD SHARING:
Plan to Share IPD: Yes
A de-identified dataset (i.e., containing no raw location/GPS information) will be generated and made available to the research community. The dataset will be stripped of all codes or any other information that could be linked back to the original data or to an individual participant. Prospective users of this dataset must agree to a confidentiality agreement, meaning that they must get permission from the HeartSteps Primary Investigator to share the data with anyone else. All external requests for data will be directed to Dr. Predrag Klasnja. Prospective investigators will submit a written proposal to the HeartSteps Investigator Team outlining the question they will investigate, the specific variables that they need to answer that question, their analytic plan for answering that question, and documentation of sufficient Institutional Review Board oversight (e.g., approval or exemption). Investigators will also need to sign a confidentiality agreement.
Supporting Information: Study Protocol

REFERENCES:
- [Background] Boruvka A, Almirall D, Witkiewitz K, Murphy SA. Assessing Time-Varying Causal Effect Moderation in Mobile Health. J Am Stat Assoc. 2018;113(523):1112-1121. doi: 10.1080/01621459.2017.1305274. Epub 2017 Mar 29. PMID 30467446
- [Background] Klasnja P, Hekler EB, Shiffman S, Boruvka A, Almirall D, Tewari A, Murphy SA. Microrandomized trials: An experimental design for developing just-in-time adaptive interventions. Health Psychol. 2015 Dec;34S(0):1220-8. doi: 10.1037/hea0000305. PMID 26651463
- [Background] Liao P, Klasnja P, Tewari A, Murphy SA. Sample size calculations for micro-randomized trials in mHealth. Stat Med. 2016 May 30;35(12):1944-71. doi: 10.1002/sim.6847. Epub 2015 Dec 28. PMID 26707831
- [Derived] Klasnja P, Smith S, Seewald NJ, Lee A, Hall K, Luers B, Hekler EB, Murphy SA. Efficacy of Contextually Tailored Suggestions for Physical Activity: A Micro-randomized Optimization Trial of HeartSteps. Ann Behav Med. 2019 May 3;53(6):573-582. doi: 10.1093/abm/kay067. PMID 30192907